CLINICAL TRIAL: NCT02894021
Title: PREvention of Post-mastectomy LYMphoceles by PAdding. A Randomized Prospective Multicenter Study
Brief Title: PREvention of Post-mastectomy LYMphoceles by PAdding
Acronym: PRELYMCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2013_843_0001
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Mastectomy
Keywords: padding; lymphoceles; prevention
MeSH Terms: conditions — Lymphocele

ARMS (2):
- classic closure (Active Comparator): mastectomy with classic closure in 2 steps, drainage by negative pressure aspiration
  Interventions: Procedure: classic closure
- padding (Experimental): areas of padding and stiching between subcutaneous tissue and pectoral muscle followed by closure in 2 steps, drainage by negative pressure aspiration for 48 h.
  Interventions: Procedure: padding

INTERVENTIONS:
Procedure: classic closure — mastectomy with classic closure in 2 steps, drainage by negative pressure aspiration
  Arms: classic closure
Procedure: padding — areas of padding and running sutures between subcutaneous tissue and pectoral muscle followed by closure in 2 steps, drainage by negative pressure aspiration for 48 h
  Arms: padding

SUMMARY:
Lymphoceles, or seromas, are the most frequent complication following mastectomy and are associated or not with axillary dissection occurring in 10 to 90% of cases. It is defined as the presence of a palpable post operative serous accumulation that is bothersome for the patient and requires a puncture and drainage or even several repeated punctures. The presence of seromas is therefore associated with discomfort and pain. Seromas could also be responsible for increased morbidity due to complications such as infection, suture separating, lymphedema, prolonged of hospital stay, or a delay in initiation of adjunct treatment (e.g. chemotherapy, radiotherapy). Some risk factors have been identified, such as obesity, increased post operative drainage of J1 to J3, and arterial hypertension.

Different measures have demonstrated the benefits of limiting axillary lymphoceles after dissection : placement of a drain, padding and delay in shoulder mobility.

Studies have shown that axillary padding decreases lymphocele development and shortens the length of hospital stay. Some studies based on padding of the mastectomy site also have shown a decrease in post operative seromas; however no study has been done on the usefulness of padding in the mastectomy site alone because they include both padding and a drain or padding of the axillary area.

The padding technique the investigators employ is performed at the donor site in breast reconstruction by latissimus dorsi muscle flap, demonstrating a reduction in the rate of seromas.

In this study, the classic technique will be compared to padding in the mastectomy site with short drainage (48h).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Female gender
* Patients with infiltrating or in situ breast cancer
* Indication of surgical treatment by mastectomy
* Patient providing written informed consent
* Patient with health insurance coverage
* Ability to provide voluntary written informed consent

Exclusion Criteria:

* Informed consent cannot be obtain
* Pregnant or lactating women
* Patients undergoing immediate breast reconstruction
* Patients with cancer untreatable by mastectomy, non curative mastectomy: partial mastectomies, preventive mastectomies (BRCA genetic mutations)
* Patients under legal protection or unable to come to a center
* Patients unable to express voluntary consent
* Patients receiving post operative anticoagulants or platelet antiaggregants
* Patients requiring postoperative anticoagulants
* Bilateral mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
postoperative lymphoceles | Day 15
  presence or absence of postoperative lymphoceles

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - CH Compiègne, Compiègne
  - CH Soissons, Soissons